CLINICAL TRIAL: NCT00562848
Title: A First-Time-in-Human Randomized Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Escalating Doses of the Oral Motilin Receptor Agonist GSK962040, in Male and Female Healthy Subjects
Brief Title: A Study to Evaluate Safety, Side Effects, Muscle Activity and Speed of Gastric Emptying of GSK962040
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: MOT107043
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Gastroparesis
Keywords: gastric emptying; pharmacokinetic; tolerability; safety; GSK962040; gut motility; First Time in Human
MeSH Terms: conditions — Gastroparesis | interventions — N-(3-fluorophenyl)-1-((4-(((3S)-3-methyl-1-piperazinyl)methyl)phenyl)acetyl)-4-piperidinamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subjects enrolled in single dose escalation cohort (Experimental): Subjects will receive escalated doses of GSK962040 with a starting dose of 1 milligrams along with placebo in fasted state.
  Interventions: Drug: GSK962040; Drug: Placebo
- Subjects enrolled in gastric emptying cohort (Experimental): Subjects will receive escalated doses of GSK962040 with a starting dose of 1 milligrams along with placebo in fasted state.
  Interventions: Drug: GSK962040; Drug: Placebo
- Subjects enrolled in gastro-enteral contractility cohort (Experimental): Eligible subjects will receive GSK962040 and placebo in the fasted state in crossover manner.
  Interventions: Drug: GSK962040; Drug: Placebo

INTERVENTIONS:
Drug: GSK962040 — GSK962040 will be supplied in the following tablet strengths: 1 milligram, 5m milligrams, 25 milligrams, 125 milligrams.
Drug: Placebo — Subjects will receive placebo.

SUMMARY:
Motilin is a peptide whose action is controlled by motilin receptors located in the gut. Action of Motilin at motilin receptors increases the gastric emptying rate (rate of emptying of food and fluid from the stomach). Compounds which stimulate motilin receptors therefore provide a potential approach to the treatment of a range of clinical conditions where delayed gastric emptying may contribute to symptoms, such as enteral feeding intolerance (post-operative or intensive care patients), gastroparesis, diabetic gastroparesis, and functional dyspepsia.

This study is the First Time In Human study for the motilin receptor agonist, GSK962040.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged between 18 and 55 years inclusive. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history (including family), physical examination, laboratory studies, and other tests.

A female subject may be enrolled in the study regardless of whether she is currently of non-childbearing potential or of childbearing potential, as long as the following conditions are observed:

- Females of non-childbearing potential: These are defined as females, regardless of their age, with functioning ovaries and who have a current documented tubal ligation [Hatcher, 2004] or hysterectomy, or females who are post-menopausal.

- Females of childbearing potential: These are defined as females, regardless of their age, with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility. This category includes females with oligomenorrhea and females who are perimenopausal.

To be eligible for the study, the female of childbearing potential

* must have a negative pregnancy test at screening before enrolment into the study; and
* must agree to use one of the highly effective methods for avoiding pregnancy in the protocol, from the Screening Visit throughout the duration of the study up to and including the follow-up clinic visit, which is anticipated to take place 7-10 days after the last dose of study medication (however the timing of the follow-up visit may be adjusted by File Note if it is indicated from the interim PK analyses). At this stage of development, there is no information on the potential pharmacokinetic interaction between GSK962040 and hormonal birth control methods, so the hormonal methods will not be acceptable.

  * A 12-lead ECG at pre-study screening, which in the opinion of the Principal Investigator or physician designee has no abnormalities that will compromise safety in this study. QT/QTc criteria are defined in the protocol.
  * A 24h Holter ECG at pre-study screening which in the opinion of the Principal Investigator or physician designee has no abnormalities that will compromise safety in this study.
  * Normal physical examination (physical exam demonstrates no evidence of clinically active disease or physical or mental impairment).
  * No abnormality on relevant clinical chemistry or haematology examination at the pre-study medical examination.
  * Body weight ≥50 kg and BMI within the range 18.5-29.9 kg/m2 inclusive where BMI = Weight in kg (height in meters)2
  * The volunteer is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
  * Signed and dated written informed consent prior to the performance of any study related procedure.
  * Subjects will have negative Helicobacter pylori status or have received eradication within the last calendar year.

Exclusion Criteria:

* Use of any hormonal method of contraception or any form of HRT (female subjects only).
* History or presence of any clinically significant metabolic, gastrointestinal or endocrinological condition.
* History or presence of clinically significant gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of major gastrointestinal surgical procedure within the last 10 years.
* History of cholecystectomy or biliary tract disease.
* History of immediate or delayed hypersensitivity reaction or idiosyncrasy to any drug, or other allergy that, in the opinion of the Principal Investigator or physician designee, contraindicates the subject's participation in the study. Additionally subjects with a known latex allergy should not be enrolled in C3.
* History or presence of corrected thyroid dysfunction (NOTE: subjects with hypothyroidism on a stable dose of thyroid replacement therapy are not eligible).
* Abnormal TSH or free T4 at screening/baseline.
* Unwillingness to commit to avoid excessive exposure to sunlight (or exposure whilst on a tanning bed) which would cause a sunburn reaction from Day -1 up to and including the follow-up visit.
* A positive pre-study HIV, Hepatitis B surface antigen or positive Hepatitis C antibody result at screening.
* History or presence of abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units.
* History or presence of recreational drug abuse or dependence.
* The subject has a positive pre-dose urine drug or alcohol breath test. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* If the subject is a tobacco smoker: An unwillingness to commit to stable and moderate use (as determined by the Investigator) of tobacco or nicotine-containing products, including nicotine patches/gum, during the course of the study.
* Consumption of grapefruit juice or grapefruit within 7 days prior to the first dose of study medication until the follow-up visit.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 3 weeks prior to the first dose of study medication until final evaluation, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Has received an investigational drug or has participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in study would result in donation of blood in excess of 500 ml within a 56 day period.
* For male volunteers: An unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first dose of study medication until 90 days following administration of the last dose of study medication.
* History of or current lactose intolerance.
* Women who are pregnant or breast-feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-09-10 (Actual); Primary Completion 2008-06-27 (Actual); Study Completion 2008-06-27 (Actual)

PRIMARY OUTCOMES:
Adverse Events - | for 5 days
Gastrointestinal symptoms - | for 6 hours
Blood pressure, heart rate, electrocardiography - | for 48 hours
Clinical chemistry/haematology - | for 5 days
Plasma pharmacokinetic parameters - | for 5 days

SECONDARY OUTCOMES:
Measurement of gastric emptying for 4.5 hours post-dose | 4.5 hours post-dose
Measurement of stomach muscle activity for 24 hours post-dose | 24 hours post-dose
Measurement of plasma pharmacokinetic and other blood tests for 3.5 hours post-dose | 3.5 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Deloose E, Depoortere I, de Hoon J, Van Hecken A, Dewit OE, Vasist Johnson LS, Barton ME, Dukes GE, Tack J. Manometric evaluation of the motilin receptor agonist camicinal (GSK962040) in humans. Neurogastroenterol Motil. 2018 Jan;30(1). doi: 10.1111/nmo.13173. Epub 2017 Aug 6. PMID 28782145
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study MOT107043 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MOT107043?search=study&study_ids=MOT107043#rs
- Available data/document: Statistical Analysis Plan: MOT107043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MOT107043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MOT107043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MOT107043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MOT107043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MOT107043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MOT107043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register